CLINICAL TRIAL: NCT03670901
Title: A Multinational, Randomized, Double-blind, Positive-controlled, Parallel Study to Compare the Efficacy and Safety of JHL1101 in Combination With CHOP (J-CHOP) Versus Rituximab in Combination With CHOP (R-CHOP) in Patients With Previously Untreated Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Study to Compare the Efficacy and Safety of JHL1101 Versus Rituximab in Patients With Previously Untreated Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development was stopped due to company's strategy consideration
Sponsor: JHL Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JHL-CLIN-1101-03
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JHL1101 (Experimental): 375 mg/m2 of JHL1101 is given intravenously on D1 of each cycle
  Interventions: Biological: JHL1101
- MabThera (Active Comparator): 375 mg/m2 of Rituximab is given intravenously on D1 of each cycle
  Interventions: Biological: MabThera

INTERVENTIONS:
Biological: JHL1101 — JHL1101, 100mg/10mL
  Arms: JHL1101
Biological: MabThera — Rituximab, 100mg/10mL
  Arms: MabThera

SUMMARY:
Approximately 500 subjects will be enrolled in this study. Subjects who meet the inclusion criteria will be randomized (1:1) into two groups. The study group will receive JHL1101 in combination with CHOP regimen, and the control group will receive rituximab (MabThera) in combination with CHOP. The dose of 375 mg/m2 is given intravenously on Day 1 (D1) of each cycle, and CHOP regimen is administered after the infusion of JHL1101 or rituximab is completed. Efficacy evaluation will be performed at baseline, after 3 cycles treatment (D18± 2 of Cycle 3, before the next cycle of treatment) and after 6 cycles treatment (D21±3 of Cycle 6). Subjects evaluated as progressive disease (PD) should be withdrawn from the study treatment and their subsequent treatments will be determined by the investigator. The analysis of primary endpoint is the ORR over the 6-cycle treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated patients histopathologically or cytologically diagnosed with CD20-positive DLBCL;
2. Aged ≥ 18 years and and ≤ 70 years of any gender;
3. International Prognostic Index (IPI) for Lymphoma score of 0 - 2 points;
4. Informed consent form has been signed before any specific study procedure is performed;
5. At least one measurable lesion. Intranoal lesions are defined as: the long diameter is ≥ 1.5 cm and the short diameter is ≥ 1.0 cm; for extranodal lesions, the long diameter should be ≥ 1.0 cm;
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 - 2;
7. The left ventricular ejection fraction (LVEF) measured by echocardiography is ≥ 50%;
8. The patients have sufficient organ function, including:

   * Absolute neutrophil count ≥ 15,000/ul; hemoglobin ≥ 80 g/L, platelet counts ≥ 75,000/uL;
   * Total bilirubin level ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN;
   * Serum creatinine level ≤ 1.5 × ULN;
   * Prothrombin time (PT) or activated partial thromboplastin time (APTT) or international normalized ratio (INR) ≤ 1.5 × ULN in the absence of anticoagulant therapy;
9. Men and women of childbearing age who have not undergone sterilization surgery must agree to practice effective contraception during the treatment period and within 12 months after the last administration of the study drug;
10. Have an expected survival of at least 6 months as judged by the investigator.

Exclusion Criteria:

1. Participated in other interventional clinical trials within three months prior to enrollment. Patients participating in non-interventional trials are eligible to participate in this study;
2. Have received blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colonystimulating factor (GM-CSF) for treatment within 14 days before enrollment;
3. Patients who are or plan to be immunized with live virus vaccine within 28 days (or within 5 half-lives of the drug) before enrollment;
4. Patients who underwent or plan to undergo major surgery within 28 days before enrollment, or patients whose surgical wounds have not healed;
5. Patients who are receiving continuous corticosteroid treatment, with > 30 mg/day prednisone or equivalent dose of corticosteroids for ≥ 10 days of continuous treatment;
6. Have a history of gastrointestinal perforation and/or fistula within 6 months before enrollment;
7. Known to be allergic to monoclonal antibody (mAb) therapy or rituximab,or patients with known sensitivity or allergy to murine products;
8. Patients who have contraindications to any component of the CHOP regimen;
9. Have previously received treatment for DLBCL, including:

   chemotherapy, immunotherapy, local radiotherapy for lymphoma, surgical treatment (except for tumor or pathologic biopsy and surgical resection not for lymphoma), and any monoclonal antibody therapy within 3 months prior to enrollment;
10. Have previously received cytotoxic drugs or anti-CD20 monoclonal antibody therapy for other diseases (such as rheumatoid arthritis);
11. Have a history of other malignancies that may affect study protocol compliance or result analysis;
12. Also suffering from severe non-malignant diseases that can affect study protocol compliance, such as severe cardiovascular diseases, uncontrolled diabetes and hypertension, peripheral nervous system or central nervous system diseases;
13. Known to have uncontrollable active infectious diseases or any major infection events (other than neoplastic fever) requiring intravenous antibiotic treatment or hospitalization within four weeks prior to enrollment;
14. Subjects known to be positive for human immunodeficiency virus (HIV) antibody;
15. Positive for hepatitis C virus (HCV) antigen or antibody;
16. Patients with HBs Ag(＋), and his/her HBV-DNA level is>103 copies;
17. The investigator believes the subject is unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 18 weeks
  To compare the overall response rate after 6 cycles treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD/PhD, Principal Investigator — Beijing Cancer Hospital, China
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No